CLINICAL TRIAL: NCT04617938
Title: Development and Implementation of a Culturally Centered Opioid Prevention Intervention for American Indian/Alaska Native Young Adults in California
Brief Title: TACUNA (Traditions and Connections for Urban Native Americans)
Acronym: TACUNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of California, Los Angeles (Other); Sacred Path Indigenous Wellness Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4UH3DA050235 (NIH)
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use; Alcohol Drinking; Marijuana Use
Keywords: American Indian/Alaska Native young adults; Cultural intervention; Motivational interviewing
MeSH Terms: conditions — Alcohol Drinking; Marijuana Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACUNA (Experimental): Randomized participants will attend 3 virtual TACUNA workshops, focused on behavioral, physical, and spiritual domains, and designed to guide AI/AN youth to make healthy choices surrounding opioid and AOD use. They will also attend a Wellness Circle, focused on healthy social networks and engaging in traditional practices.
  Interventions: Behavioral: TACUNA plus Wellness Circle
- Opioid education (Active Comparator): Randomized participants will attend 1 virtual opioid education workshop, focused on behavioral and physical domains, and designed to guide AI/AN youth to make healthy choices surrounding opioid and AOD use.
  Interventions: Behavioral: Opioid Education Workshop

INTERVENTIONS:
Behavioral: TACUNA plus Wellness Circle — TACUNA provides three virtual workshops (one hour each) that use motivational interviewing and a virtual Wellness Circle (WC). The workshops combine a 30-minute discussion of opioid, alcohol and marijuana use, and social networks with another 30 minutes focused on three different traditional practices (one per workshop). TACUNA was adapted from our three-session workshop, MICUNAY (Motivational Interviewing and Culture for Urban Native American Youth) protocol, which was developed and tested for urban AI/AN adolescents and from focus groups conducted in Year 1. For the Wellness Circle, youth will have members of their social network virtually attend these once-a-month gatherings. The WC will bring people together to celebrate health and wellness and tradition. The WC will focus on the importance of social networks in making healthy choices, and provide discussion on the role that AOD use and engagement in traditional practices among members of their social networks affect their choices.
  Arms: TACUNA
Behavioral: Opioid Education Workshop — The virtual opioid education workshop draws from prevention and education materials supplied and recommended by the National AI/AN Technology and Transfer Center, which is funded by SAMHSA. Materials are culturally relevant educational packages addressing opioid use through recorded webinars, toolkits, and other resources.
  Arms: Opioid education

SUMMARY:
This study responds to Request For Application-DA-19-035, HEAL (Helping End Addiction Long Term) initiative: Preventing OUD in Older Adolescents and Young Adults (ages 16-30) by developing and implementing a culturally centered intervention to address opioid use among urban AI/AN emerging adults in California. The primary goal of this study is to compare AI/AN emerging adults who receive TACUNA plus a Wellness Circle (WC) to those AI/AN emerging adults who receive an opioid education workshop on outcomes (e.g., opioid misuse and alcohol and other drug use) over a period of 12 months. TACUNA will be a motivational interviewing group intervention that incorporates traditional practices and discussion of how to cultivate healthy social networks and cultural worlds. The Wellness gathering will be for emerging adults and people in their social network, and will focus on how social networks and cultural connectedness influence healthy behaviors. Opioid education will focus on discussion of opioid misuse within the AI/AN urban community and ways to reduce use in a culturally appropriate manner. Investigators expect those who receive TACUNA + WG will report less opioid and AOD (alcohol and other drug) use frequency, fewer consequences, less time spent around peers who use opioids and AOD, and less perceived prevalence of peer use compared to opioid education over a period of 12 months. Also, investigators will evaluate the intervention's effects on secondary outcomes of social networks and cultural connectedness. Survey data is collected at baseline, 3-months, 6-months and 12-months. Longitudinal analyses will compare intervention participant and control participants on primary and secondary outcomes.

DETAILED DESCRIPTION:
Data from 2015 show that American Indians/Alaska Natives (AI/ANs) have the highest rates of diagnosis for opioid use disorders (OUD) and deaths from drug overdose. Misuse of prescription opioids, defined here as taking opioid medications in a manner or dose other than prescribed or for hedonic effects, and the use of heroin, have emerged as major public health concerns in the United States. Of particular concern is the prevalence of opioid use among emerging adults (ages 18-25) as this is a developmental period of heightened vulnerability and critical social, neurological, and psychological development.

Unique risk factors may predispose urban AI/AN young adults to use opioids, alcohol or other drugs. For example, experiences of acculturative stress directly and indirectly associated with historical trauma experienced by AI/ANs throughout U.S. history result in poor health outcomes. One U.S. law that has been postulated to contribute to various health disparities among urban AI/ANs is the Relocation Act of 1956. This Act financed the relocation of individual AIs and AI families to job training centers in designated U.S. cities. Rather than establishing economic stability, large numbers of AIs who moved to urban areas became unemployed, homeless, and disconnected from their community-based support networks. This relocation appears to have contributed to an inter-generational effect whereby successive generations of urban AIs and ANs continue to experience various health-related disparities. Our work with urban AI/AN adolescents highlighted that many experience stress related to identity in the form of both subtle (e.g., being asked whether one is a "real" Indian) and overt (e.g., being called a racist name like Squaw or Red Skin) discrimination. Programming that incorporates traditional practices, promotes community involvement, and encourages healthy notions of AI/AN identity may increase well-being and healthy behaviors by addressing sources of stress linked to cultural identity, stigma, and community connections. However, few evidence-based programs that integrate these cultural elements have been developed, implemented, and evaluated with urban AI/AN using a strong research design. The current study substantially extends work with AI/AN emerging adults by adapting and testing an integrated culturally appropriate MI and social network intervention to address opioid and other AOD (alcohol and other drug) misuse at both the individual and community level.

ELIGIBILITY:
Inclusion Criteria:

* must self-identify as American Indian/Alaska Native (AI/AN)
* be in the age range of 18-25
* not be in need of substance treatment

Exclusion Criteria:

* If substance treatment need is indicated

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 541 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Frequency of opioid use | change from baseline to 3 months
  We will assess frequency of opioid use in the past three months from 1 = never to 6 = over 20 times.
Frequency of opioid use | change from baseline to 6 months
  We will assess frequency of opioid use in the past three months from 1 = never to 6 = over 20 times.
Frequency of opioid use | change from baseline to 12 months
  We will assess frequency of opioid use in the past three months from 1 = never to 6 = over 20 times.
Frequency of alcohol and marijuana use | change from baseline to 3 months
  We will assess frequency of alcohol and marijuana use in the past three months from 1 = never to 6 = over 20 times.
Frequency of alcohol and marijuana use | change from baseline to 6 months
  We will assess frequency of alcohol and marijuana use in the past three months from 1 = never to 6 = over 20 times.
Frequency of alcohol and marijuana use | change from baseline to 12 months
  We will assess frequency of alcohol and marijuana use in the past three months from 1 = never to 6 = over 20 times.

SECONDARY OUTCOMES:
Network Composition | change from baseline to 3 months
  Participants will be asked to name 15 contacts ("alters") who are at least 18 years of age. Participants will rate each of the 15 people on the same set of questions with categorical response options (about demographics, relationship quality, likelihood to use drugs, etc.). For each participants the selected responses will be summed across all of the network alters and divided by 15 to produce network composition percentages of the whole set of alters named by the participant (% of AI/Ans, % who engage in heavy drinking).
Network Composition | change from baseline to 6 months
  Participants will be asked to name 15 contacts ("alters") who are at least 18 years of age. Participants will rate each of the 15 people on the same set of questions with categorical response options (about demographics, relationship quality, likelihood to use drugs, etc.). For each participants the selected responses will be summed across all of the network alters and divided by 15 to produce network composition percentages of the whole set of alters named by the participant (% of AI/Ans, % who engage in heavy drinking).
Network Composition | change from baseline to 12 months
  Participants will be asked to name 15 contacts ("alters") who are at least 18 years of age. Participants will rate each of the 15 people on the same set of questions with categorical response options (about demographics, relationship quality, likelihood to use drugs, etc.). For each participants the selected responses will be summed across all of the network alters and divided by 15 to produce network composition percentages of the whole set of alters named by the participant (% of AI/Ans, % who engage in heavy drinking).
Cultural connectedness | change from baseline to 3 months
  Cultural connectedness will be measured with 29 items that address 3 dimensions: identity, traditions, and spirituality. Respondents answer 11 yes/no questions (e.g., I have a traditional person, Elder, or other person who I talk to), and use a scale from 1= "strongly disagree" to 5= "strongly agree" for 18 items (e.g., I feel a strong connection/attachment towards my Native American community or Tribe).
Cultural connectedness | change from baseline to 6 months
  Cultural connectedness will be measured with 29 items that address 3 dimensions: identity, traditions, and spirituality. Respondents answer 11 yes/no questions (e.g., I have a traditional person, Elder, or other person who I talk to), and use a scale from 1= "strongly disagree" to 5= "strongly agree" for 18 items (e.g., I feel a strong connection/attachment towards my Native American community or Tribe).
Cultural connectedness | change from baseline to 12 months
  Cultural connectedness will be measured with 29 items that address 3 dimensions: identity, traditions, and spirituality. Respondents answer 11 yes/no questions (e.g., I have a traditional person, Elder, or other person who I talk to), and use a scale from 1= "strongly disagree" to 5= "strongly agree" for 18 items (e.g., I feel a strong connection/attachment towards my Native American community or Tribe).
Network Structure | change from baseline to 3 months
  Participants will rate the relationship strength between each of the 15 named alters. For each alter pair they will rate if the two people know each other and, if yes, have they connected recently. Measures of network structure (i.e. network "connectedness") will be constructed from the set of evaluations for each participant. For example, network "density" will be constructed for the network overall, which is calculated by summing the number of alter pairs who know each other and dividing by the total number of possible ties among 15 alters (105). Individual alter "centrality" will be calculated by summing the number of connections each individual alter has with other alters in the network.
Network Structure | change from baseline to 6 months
  Participants will rate the relationship strength between each of the 15 named alters. For each alter pair they will rate if the two people know each other and, if yes, have they connected recently. Measures of network structure (i.e. network "connectedness") will be constructed from the set of evaluations for each participant. For example, network "density" will be constructed for the network overall, which is calculated by summing the number of alter pairs who know each other and dividing by the total number of possible ties among 15 alters (105). Individual alter "centrality" will be calculated by summing the number of connections each individual alter has with other alters in the network.
Network Structure | change from baseline to 12 months
  Participants will rate the relationship strength between each of the 15 named alters. For each alter pair they will rate if the two people know each other and, if yes, have they connected recently. Measures of network structure (i.e. network "connectedness") will be constructed from the set of evaluations for each participant. For example, network "density" will be constructed for the network overall, which is calculated by summing the number of alter pairs who know each other and dividing by the total number of possible ties among 15 alters (105). Individual alter "centrality" will be calculated by summing the number of connections each individual alter has with other alters in the network.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth D'Amico, PhD, Principal Investigator — RAND; Daniel Dickerson, DO, MPH, Principal Investigator — UCLA Integrated Substance Abuse Programs
Locations (3):
- United States (3):
  - United American Indian Involvement, Inc, Los Angeles, California
  - UCLA, Los Angeles, California
  - RAND Corporation, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuklinski MR, Gibbons BJ, Bowser DM, McCollister KE, Smart R, Dunlap LJ, Shenkar E, Bonar EE, Boomer T, Campbell M, Fiellin LE, Hutton DW, Rao V, Saldana L, Su K, Walton MA, Yilmazer T. Investing in Interventions to Prevent Opioid Use Disorder in Adolescents and Young Adults: Start-up Costs from NIDA's HEAL Prevention Initiative. Prev Sci. 2025 Nov;26(7):1045-1055. doi: 10.1007/s11121-025-01835-6. Epub 2025 Oct 14. PMID 41085955
- [Derived] D'Amico EJ, Kennedy DP, Malika N, Klein DJ, Brown RA, Rodriguez A, Johnson CL, Schweigman K, Arvizu-Sanchez V, Etz K, Dickerson DL. Risk and protective factors of social networks on alcohol, cannabis, and opioid use among urban American Indian/Alaska Native emerging adults. Psychol Addict Behav. 2023 Aug;37(5):657-669. doi: 10.1037/adb0000918. Epub 2023 Apr 6. PMID 37023284
- [Derived] Kennedy DP, D'Amico EJ, Brown RA, Palimaru AI, Dickerson DL, Johnson CL, Lopez A. Feasibility and acceptability of incorporating social network visualizations into a culturally centered motivational network intervention to prevent substance use among urban Native American emerging adults: a qualitative study. Addict Sci Clin Pract. 2022 Sep 30;17(1):53. doi: 10.1186/s13722-022-00334-1. PMID 36180896
- [Derived] D'Amico EJ, Dickerson DL, Rodriguez A, Brown RA, Kennedy DP, Palimaru AI, Johnson C, Smart R, Klein DJ, Parker J, McDonald K, Woodward MJ, Gudgell N. Integrating traditional practices and social network visualization to prevent substance use: study protocol for a randomized controlled trial among urban Native American emerging adults. Addict Sci Clin Pract. 2021 Sep 26;16(1):56. doi: 10.1186/s13722-021-00265-3. PMID 34565444

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04617938/Prot_SAP_002.pdf
  • Informed Consent Form (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT04617938/ICF_000.pdf